CLINICAL TRIAL: NCT06569862
Title: Comparison of the Risk of Surgical Site Infections Between Dressings Stopped at Postoperative Day 1 vs Dressings Stopped at Postoperative Day 6+/-1 After Elective Abdominal Surgery: a Multicentre Non-inferiority Randomized Controlled Trial
Brief Title: Comparison of the Risk of Surgical Site Infections Between Dressings Stopped at Postoperative Day 1 vs Dressings Stopped at Postoperative Day 6+/-1 After Elective Abdominal Surgery
Acronym: PAN-STOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: APHP230859
Record Dates: First submitted 2024-06-28; First posted 2024-08-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Elective Abdominal Surgery
Keywords: Surgical site infection; Dressing; Elective abdominal surgery; Postoperative care
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative day 1 dressing (Experimental): After removing the dressing on day 1, no dressing change by a nurse is required.
  Interventions: Procedure: Postoperative day 1 dressing
- Postoperative day 6+/-1 dressing (Other): Daily dressing changes should be performed according to standard nursing procedures until postoperative day 6 (+/-1)
  Interventions: Procedure: Postoperative day 6+/-1 dressing

INTERVENTIONS:
Procedure: Postoperative day 1 dressing — The patient's dressing will be removed on the first day after surgery, leaving the incision exposed to air, with daily cleaning.
  Arms: Postoperative day 1 dressing
Procedure: Postoperative day 6+/-1 dressing — The patient will have a daily dressing change according to the usual nursing procedures, including saline serum washing, until the sixth day (+/- 1 day) after surgery. This will be done while the patient is in hospital, or at home if discharged before the sixth day.
  Arms: Postoperative day 6+/-1 dressing

SUMMARY:
The daily changing of postoperative dressings is a widespread practice, often continuing until the 5th-7th day after surgery. In theory, dressings aim to reduce the risk of superficial surgical site infections (SSIs). However, several studies have suggested that early removal of the dressing does not significantly impact the rate of superficial SSIs, and this approach is now applied in clinical practice by several teams. A Cochrane review indicated that the absence of dressing does not appear to be harmful, though it emphasized the very low level of evidence provided and the need for high-quality randomized controlled trials. In this study, the investigators aim to provide high-level evidence on the effect of stopping dressings from the 1st postoperative day and the lack of impact on the risk of SSIs, to standardize practices and enable recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age (≥18 years)
* Scheduled for elective abdominal surgery requiring a skin incision of at least 4 cm long listed below:

All pancreatectomies, All hepatectomies, All splenectomies, All adrenalectomies, All bariatric surgeries, All gastric surgeries, including gastrectomy and reflux surgery, All parietal surgeries; ventral hernia repairs, inguinal or femoral hernia repairs, with or without mesh placement..

All small bowel resections, Laparotomy cholecystectomies, All duodenal surgeries, Right, transverse or left colectomy, by laparotomy or laparoscopy, provided that there is a skin incision for extraction of the surgical specimen, but without the presence or creation of a stoma Proctectomy but without the presence or creation of a stoma

* Class I or II (clean or clean-contaminated) according to the ALTEMEIER classification
* Affiliated in a Social Security scheme (beneficiary or entitled person, excluding AME)
* Have signed an informed consent form

Exclusion Criteria:

* Presence or completion of a stoma
* Previous abdominal surgery in the month prior to inclusion
* Emergency surgery
* Outpatient surgery
* Closure by biological glue
* Active bacterial infection at the time of surgery or recent antibiotic therapy (up to 15 days before surgery)
* Neutrophil count < 500/mm3 at time of surgery
* Grade B or C cirrhosis (Child-Pugh classification)
* Pregnancy
* Breast-feeding
* Patient under guardianship or curatorship
* Patient deprived of liberty by judicial or administrative decision
* Patient unable to perform perioperative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1288 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of superficial surgical site infections (SSI) | Day 30 post-surgery
  The percentage of superficial surgical site infections (SSI) within the 30 days following surgery, defined according to the criteria set by the Centers for Disease Control and Prevention (CDC).

SECONDARY OUTCOMES:
Direct and indirect costs | Day 30 post-surgery
  Medical-economic impact
Rate of repeat surgery | 30 days post-surgery
Rate of unscheduled nursing care | 30 days post-surgery
Percentage of patients who asked for their scars to be covered | 30 days post-surgery
Total length of hospital stay | 30 days post-surgery
Overall morbidity rate according to Clavien-Dindo | 30 days post-surgery
Rate of antibiotic treatment | 30 days post-surgery
Quality of life for patients | Day 6 and Day 30 post-surgery
  Patient's quality of life on days 6 and 30 post-surgery as assessed using the EuroQol Research Foundation 5 Dimensions Self-Questionnaire (EQ-5D-5L).
The incremental cost-effectiveness ratio (ICER) | 30 days after inclusion
  The incremental cost-effectiveness ratio (ICER) measures the costs (from the healthcare system perspective) per infection prevented between the intervention and control arms 30 days after inclusion. It is calculated as the difference in average costs between the two arms divided by the difference in average number of infections between them.
The incremental cost-utility ratio (ICUR) | 30 days after inclusion
  The incremental cost-utility ratio (ICUR) assesses the costs (from the healthcare system perspective) per Quality-Adjusted Life Year (QALY) gained between the intervention arm and the control arm 30 days after inclusion. Quality of life is evaluated using the EQ-5D-5L scale (EuroQol Group) at the inclusion visit, discharge from hospital, and at 30 days, covering five dimensions (mobility, stress/anxiety, ability to perform daily activities, autonomy, pain/discomfort). ICUR is calculated as the difference in average costs between the two arms divided by the difference in average QALYs gained between them.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Pitié-Salpêtriere - APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.